CLINICAL TRIAL: NCT01372332
Title: Assessment of Homonymous Visual Loss and Its Impact on Visual Exploration, Activities of Daily Living (ADL) and Quality of Life (QoL)
Acronym: Hemi-Drive
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ulrich Schiefer, Prof. Dr. med., University Hospital Tuebingen
Other Study IDs: 086/2011BO2
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Homonymous Hemianopia
Keywords: homonymous hemianopia; quality of life (QoL); visual exploration; on-road car driving; driving simulator; useful field of view (UFOV); modified field of view (MAFOV)
MeSH Terms: conditions — Hemianopsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal subjects: Age-related (+ 5 years of age) and gender-matched normal subjects.
- Patients with homonymous hemianopia: Patients with homonymous visual field defects

SUMMARY:
The purpose of this explorative study, targeting subjects with homonymous visual field loss, is threefold:

(i) to identify the perimetric / psychophysical method, that is most closely correlated with an individually assessed quality of life (QoL) score, using a validated questionnaire (NEI-VFQ 25) (ii) to determine, whether gaze-related (exploratory eye movements) or visual field-related (eyes steadily fixating) parameters are better for the characterization of the visual capacities that are necessary for activities of daily living (ADL), as represented by (iia) a standardized visual search task ("supermarket special offer search task") (iib) by an on-road car driving pilot study.

ELIGIBILITY:
Inclusion Criteria:

- Patients with homonymous visual field defects Primary inclusion criterion: (Stable) homonymous visual field defects, as obtained by binocular semi-automated kinetic perimetry (SKP), using the III4e stimulus, within on onset of at least six months ago, due to a vascular or a traumatic lesion.

Further inclusion criteria: (i) general: physical, intellectual and linguistic abilities, necessary to understand the test requirements: no mobility limitations / hemiparesis, Minimental Status Examination Test score above 24, adequate knowledge of the German language, willingness to comply with the protocol, > 18 years, informed consent.

(ii) Ophthalmological: spherical ametropia max. ± 8 dpt, cylindrical ametropia max. ± 3 dpt, best corrected distant visual acuity > 6/12 (= 0.5), isocoria, pupil diameter > 3 mm, intraocular pressure ≤ 21 mmHg, normal anterior segments, no clinically relevant media opacities, normal appearance of the optic disc (cup to disc ratio = CDR ≤ 0.5, intraocular difference of CDR < 0.3).

- Normal subjects (i) General inclusion criteria: Physical, intellectual and linguistic abilities needed to understand the test requirements: no mobility limimtaions / hemiparesis, Minimental Status Examination Test score above 24, adequate knowledge of the German language, willingness to comply with the protocol, > 18 years, informed consent.

(ii) Ophthalmological inclusion criteria: maximum allowed spherical ametropia at distance is ± 6.00 diopters and the maximum cylindrical ametropia is ± 2 diopters. The best corrected distance visual acuities are equal to, or better than 20/20 and 1.0, respectively, for those aged up to 60 years; better than 20/25 and 0.8 for those aged between 60 and 70 years; and better than, or equal to, 20/33 and 0.6 for those aged more than 70 years. All participants manifest equal pupil size, pupil diameter > 3 mm, no relative afferent pupillary defect, intraocular pressure ≤ 21 mmHg, normal anterior segments, no clinically relevant media opacities, normal appearance of the optic disc (cup to disc ratio = CDR ≤ 0.5, intraocular difference of CDR < 0.3) and normal central and peripheral fundus findings on direct and indirect undilated ophthalmoscopic examination.

Exclusion Criteria:

- Patients with homonymous visual field defects: (i) General exclusion criteria: Pregnancy, nursing, asthma, HIV+ or AIDS, history of epilepsy or significant psychiatric disease, history of drug and alcohol abuse, Minimental Status Examination Test score below 24, medications known to affect visual field sensitivity.

(ii) Ophthalmological exclusion criteria: diabetic retinopathy, infections (e.g. keratitis, conjunctivitis, uveitis), severe dry eyes, miotic drug, amblyopia, squint, nystagmus, albinism, any ocular pathology, in either eye, that may interfere with the ability to obtain visual fields, disc imaging or accurate IOP readings, keratoconus, intraocular surgery (except for uncomplicated cataract surgery) performed < 3 month prior to screening, protanopia, deuteranopia, history or presence of macular disease and / or macular edema, ocular trauma.

- Normal subjects: (i) General exclusion criteria: pregnancy, nursing, mental or neurological diseases, Minimental Status Examination Test score below 24, history of coronary heart disease, stroke, diabetes mellitus, migraine, vasospasm/ Raynaud's disease, drugs indicating severe systemic diseases (e.g. anti-diabetic or anti-hypertensive medication for subjects under 70 years of age), drugs or medications influencing reaction time, history of drug and alcohol abuse, suspected lack of compliance. Subjects over 70 years of age will not be excluded for use of anti-hypertensive medication.

(ii) Ophthalmological exclusion criteria: Amblyopia, strabismus, ocular motility disorders, retinal pathology, glaucoma, suspicion of glaucoma, ocular hypertension or any other sign of other optic neuropathy, macular degeneration, protanopia, deuteranopia, eye surgery (except for uncomplicated cataract surgery), any type of refractive surgery, history or signs of neuro-ophthalmological diseases, acute infections, diabetic retinopathy, use of miotic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 patients with homonymous visual field defects and 30 age-related (+ 5 years of age) and gender-matched normal subjects. All subjects are free to stop participation of the tests at any time without any consequences on the future treatment of the patient. The circumstances of any discontinuation will be documented.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Identification of the perimetric / psychophysical method, that is most closely correlated with an individually assessed quality of life (QoL) score | 2 years
  Quality of life (QoL) is better correlated with the modified ESTERMAN score of the binocular semi-automated kinetic perimetry of the 90° visual field than with the number of affected test locations (local sensitivity < 10 dB) according to the binocular integrated visual field (IVF)

SECONDARY OUTCOMES:
Exploration whether gaze-related or visual field-related parameters are better for the characterization of the visual capacities that are necessary for activities of daily living (ADL) | 2 years
  1. Activities of daily living ("supermarket special offer search task"), are better correlated with the modified ESTERMAN score, based on the intact binocular gaze field than with the modified ESTERMAN score, based on the binocular semi-automated kinetic perimetry of the 90° visual field (90° SKP)
  2. Activities of daily living (driving performance) are better correlated with (the ESTERMAN score, based on) the intact binocular gaze field than with the UFOV risk score

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schiefer, Prof. Dr.med., Principal Investigator — Centre for Ophthalmology Institute for Ophthalmic Research University of Tübingen
Locations (1):
- Centre for Ophthalmology Institute for Ophthalmic Research University of Tübingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Kasneci E, Sippel K, Aehling K, Heister M, Rosenstiel W, Schiefer U, Papageorgiou E. Driving with binocular visual field loss? A study on a supervised on-road parcours with simultaneous eye and head tracking. PLoS One. 2014 Feb 11;9(2):e87470. doi: 10.1371/journal.pone.0087470. eCollection 2014. PMID 24523869
- [Background] Kübler T, Kasneci E, Rosenstiel W, Schiefer U, Nagel K, Papageorgiou E. Stress-indicators and exploratory gaze for the analysis of hazard perception in patients with visual field loss. Science Direct, Transportation Research Part F 24: 231-43, 2014
- [Derived] Kasneci E, Sippel K, Heister M, Aehling K, Rosenstiel W, Schiefer U, Papageorgiou E. Homonymous Visual Field Loss and Its Impact on Visual Exploration: A Supermarket Study. Transl Vis Sci Technol. 2014 Nov 3;3(6):2. doi: 10.1167/tvst.3.6.2. eCollection 2014 Oct. PMID 25374771
- [Derived] Sippel K, Kasneci E, Aehling K, Heister M, Rosenstiel W, Schiefer U, Papageorgiou E. Binocular glaucomatous visual field loss and its impact on visual exploration--a supermarket study. PLoS One. 2014 Aug 27;9(8):e106089. doi: 10.1371/journal.pone.0106089. eCollection 2014. PMID 25162522